CLINICAL TRIAL: NCT00300417
Title: A Phase I Study of the Safety and Immunogenicity of a West Nile Virus Recombinant DNA Plasmid Vaccine, VRC-WNVDNA020-00-VP, in Healthy Adult Subjects
Brief Title: Phase I Study of West Nile Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060110; 06-I-0110
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-28

CONDITIONS: West Nile Fever
Keywords: Flavivirus; Mosquito; Immunity; Preventive; West Nile Fever; West Nile Virus; Vaccine; Healthy Volunteer; HV
MeSH Terms: conditions — West Nile Fever

INTERVENTIONS:
Drug: VRC-WNVDNA020-00-VP

SUMMARY:
This study will test the safety of an experimental vaccine for preventing West Nile virus infection. The virus is spread mainly by mosquito bites. Symptoms can include high fever, headache, neck stiffness, stupor, muscle weakness, vision loss, numbness and paralysis. Rarely, infection leads to permanent nerve damage and possibly death. The vaccine used in the study is made from DNA that codes for West Nile virus proteins. Injected into a muscle, the DNA instructs the body to make a small amount of West Nile virus protein. This study will see if the body creates resistance or immunity to these proteins. Participants cannot get West Nile virus from the vaccine.

Healthy normal volunteers between 18 and 65 years of age may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood and urine tests for various infections and other medical problems. Women who are able to become pregnant are given a pregnancy test. Women who are pregnant or breastfeeding may not participate. Anyone who has received a vaccination for Yellow Fever or Japanese Encephalitis virus in the past may not participate in this research study.

Participants will receive three injections of the experimental vaccine, the first on the first study day (Day 0), the second on Day 28, and the third on Day 56. The injections are given with a device called Biojector® (Registered Trademark) 2000 that delivers the vaccine through the skin into the muscle without the use of a needle. On the day of each injection, subjects are given a diary card to take home for recording their temperature and any symptoms or side effects for 5 days. They return to the clinic 2 weeks after each injection, bringing the completed card with them at that time. In addition to the injections, subjects have the following tests and procedures during clinic visits:

* Medical history and, if needed, physical examination: Day 0 and weeks 2, 4, 6, 8, 10, 12, 24 and 32
* Vital signs and weight: Day 0 and weeks 2, 4, 6, 8, 10, 12, 24 and 32
* Lymph node exam: Day 0 and weeks 2, 4, 6, 8, 10, and 12
* Blood samples: Day 0 and weeks 2, 4, 6, 8, 10, 12, 24 and 32
* Pregnancy test (for women): Day 0 and weeks 4, 8 and 32
* Urine sample: Day 0 and weeks 2, 4, 6, 8, and 10

The blood and urine tests are for health checks. Some blood samples are also used to study the immune response to the vaccine and for gene testing.

DETAILED DESCRIPTION:
Study Design: This is a Phase I open-label study to evaluate safety, tolerability, and immunogenicity of a recombinant DNA vaccine, VRC-WNVDNA020-00-VP. The hypothesis is that this regimen will be safe for human administration and elicit a higher titer of neutralizing antibody response than a prior WNV DNA vaccine. The primary objectives are to evaluate the safety and tolerability in humans of the investigational vaccine in healthy young adults and in healthy older adults. Secondary and exploratory objectives are related to the immunogenicity of the study vaccine.

Product Description: VRC-WNVDNA020-00-VP is composed of a single closed-circular DNA plasmid that encodes the WNV viral protein precursor transmembrane (prM) and envelope (E) with a CMV/R promoter. Vaccine vials will be supplied at 4 mg/mL. Each DNA vaccination will be 1 mL of vaccine administered intramuscularly (IM) in the deltoid muscle using the Biojector 2000 Needle-Free Injection Management System (Biojector).

Subjects: A total of 30 healthy adults will be enrolled in two groups: Group 1 will be comprised of 15 healthy adults 18 to 50 years old and Group 2 will be comprised of 15 healthy adults 51 to 65 years old.

Study Plan: All subjects will receive 3 injections on the schedule shown in the schema. The protocol requires nine clinic visits and three telephone follow-up contacts.

Study Duration: 32 weeks of clinical follow up for each participant. A long-term follow-up contact at Week 52 may include interim medical history and research blood draw; or subject may opt for the long-term contact to occur by telephone, e-mail or mail for the interim medical history only.

Study Endpoints: The primary endpoint is safety and tolerability of the regimen. The secondary immunogenicity endpoints are WNV neutralizing antibody, WNV specific antibody as measured by ELISA, WNV-specific T cell responses measured by intracellular cytokine staining (ICS) assay and ELISPOT. Other immunogenicity assays through Week 32 may also be completed as exploratory evaluations, as well as from the Week 52 blood samples if collected.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. 18 to 65 years old.
2. Available for clinical follow-up through Week 32 and contact (correspondence, telephone or e-mail) or clinical visit through Week 52 of the study.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Complete an Assessment of Understanding prior to enrollment and verbalize understanding of all questions answered incorrectly.
5. Able and willing to complete the informed consent process.
6. Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.
7. Willing to donate blood for sample storage to be used for future research and genetic testing, including HLA analysis.
8. In good general health without clinically significant medical history and has satisfactorily completed screening.
9. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) less than 40 within the 28 days prior to enrollment.

   Laboratory Criteria within 28 days prior to enrollment:
10. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men.
11. White blood cell (WBC) equal to 3,300-12,000 cells/mm(3).
12. Absolute neutrophil count (ANC) within institutional normal range.
13. Total lymphocyte count greater than or equal to 800 cells/mm(3).
14. Platelets equal to 125,000 - 400,000/mm(3).
15. Alanine aminotransferase (ALT; SGPT) less than or equal to 1.25 x upper limit of normal.
16. Serum creatinine less than or equal to 1 x upper limit of normal (less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males).
17. Normal urinalysis defined as negative glucose, negative or trace protein, and no clinically significant blood in the urine.
18. Negative FDA-approved HIV blood test. [Note: Results of HIV ELISA will be documented, but a negative HIV PCR will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study.]
19. Negative hepatitis B surface antigen.
20. Negative anti-HCV and negative hepatitis C virus (HCV) PCR.

    Laboratory Criteria within 12 weeks (84 days) prior to enrollment:
21. Negative flavivirus serology (in the Focus Technologies WNV antibody ELISA assay) within 84 days prior to enrollment and no history of prior vaccination against yellow fever or Japanese encephalitis virus; and no history of prior vaccination against West Nile virus with an investigational vaccine.

    Female-Specific Criteria:
22. Negative beta-HCG pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.
23. A female participant must meet any of the following criteria:

No reproductive potential because of menopause (one year without menses) or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

or

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 32 of the study,

or

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 32 of the study by one of the following methods:

* condoms, male or female, with or without a spermicide
* diaphragm or cervical cap with spermicide
* intrauterine device
* contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive method
* male partner has previously undergone a vasectomy

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply.

Women:

1. Breast-feeding or planning to become pregnant during the 32 weeks of study participation.

   Volunteer has received any of the following substances:
2. Immunosuppressive medications, cytotoxic medications, inhaled corticosteroids, or long-acting beta-agonists within the past six months. (Note that use of corticosteroid nasal spray for allergic rhinitis, topical corticosteroids for an acute uncomplicated dermatitis, or short-acting beta-agonists in controlled asthmatics are not excluded).
3. Blood products within 120 days prior to HIV screening.
4. Immunoglobulin within 60 days prior to HIV screening.
5. Investigational research agents within 30 days prior to initial study vaccine administration.
6. Live attenuated vaccines within 30 days prior to initial study vaccine administration.
7. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration.
8. Current anti-TB prophylaxis or therapy.

   Volunteer has a history of any of the following clinically significant conditions:
9. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain.
10. Autoimmune disease or immunodeficiency.
11. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
12. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
13. History of thyroidectomy or thyroid disease that required medication within the past 12 months.
14. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years.
15. Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.
16. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
17. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
18. Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.
19. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
20. Allergic reaction to aminoglycoside antibiotics.
21. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to enrollment, a history of suicide plan or attempt.
22. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.
23. Active smoker within the past 5 years AND with 25 pack-years or greater smoking history.
24. If age 51-65 years and with 3 or more of the 5 health risk factors noted below, the subject will be excluded:

    * Current smoker (or quit smoking less than 28 days prior to enrollment)
    * BMI greater than 35
    * Fasting low density lipoprotein (LDL) greater than 159 mg/dL or fasting cholesterol greater than 239 mg/dL
    * Systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
    * Fasting blood glucose greater than 125 mg/dL

Note: The fasting blood tests require 8 hours fast prior to the blood draw. The results used for eligibility screening must be from tests completed no more than 12 weeks (84 days) prior to day of enrollment. The individual criteria for BMI (inclusion item 9), blood pressure (exclusion item 15) and smoking history (exclusion item 23) must also be met.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-03-03; Study Completion 2007-12-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). West Nile virus activity--United States, September 29-October 5, 2004. MMWR Morb Mortal Wkly Rep. 2004 Oct 8;53(39):922-3. PMID 15470326
- [Derived] Ledgerwood JE, Pierson TC, Hubka SA, Desai N, Rucker S, Gordon IJ, Enama ME, Nelson S, Nason M, Gu W, Bundrant N, Koup RA, Bailer RT, Mascola JR, Nabel GJ, Graham BS; VRC 303 Study Team. A West Nile virus DNA vaccine utilizing a modified promoter induces neutralizing antibody in younger and older healthy adults in a phase I clinical trial. J Infect Dis. 2011 May 15;203(10):1396-404. doi: 10.1093/infdis/jir054. Epub 2011 Mar 11. PMID 21398392